CLINICAL TRIAL: NCT02067767
Title: Phase 2 Multicentric Open-label Study of Switch From Abacavir/Lamivudine Fixed Dose Combination Plus Nevirapine to Abacavir/Lamivudine/Dolutegravir in Virologically Suppressed HIV-1 Infected Adults
Brief Title: Multicentric Open-label Study of Switch From Abacavir/Lamivudine Fixed Dose Combination Plus Nevirapine to Abacavir/Lamivudine/Dolutegravir in Virologically Suppressed HIV-1 Infected Adults (SWAD)
Acronym: SWAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC13_0230
Record Dates: First submitted 2014-02-18; First posted 2014-02-20 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2015-02

CONDITIONS: HIV-1 Infection
Keywords: HIV-1 infection; Nevirapine; Dolutegravir; Anti-retroviral agents
MeSH Terms: interventions — abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abacavir/Lamivudine/Dolutegravir (Experimental): Patients switched from their ongoing treatment of ABC/3TC + NVP to ABC/3TC/DTG.
  Interventions: Drug: Abacavir/Lamivudine/Dolutegravir

INTERVENTIONS:
Drug: Abacavir/Lamivudine/Dolutegravir — At Day 1 (D1):
  * group 1 will switch their ongoing treatment of ABC/3TC + NVP to ABC/3TC/DTG ;
  * group 2 will continue NVP and switch ABC/3TC to ABC/3TC/DTG for 6 days (D-5 to D0), then stop NVP from D1.

SUMMARY:
Abacavir/Lamivudine + Nevirapine (ABC/3TC + NVP) is a very effective and well tolerable regimen on the long-term. However this regimen comprises 2 pills per day. Abacavir/Lamivudine/Dolutegravir (ABC/3TC/DTG) offers simplification with a single pill per day with no food constraints, Dolutegravir (DTG) having the advantage over Nevirapine (NVP) of high potency, higher genetic barrier to resistance, with a very good safety profile. The objective of this study is to evaluate the virologic safety (maintenance of virologic suppression) after switching from ABC/3TC + NVP to ABC/3TC/DTG in 50 HIV-1 infected adults with prolonged HIV RNA suppression on ABC/3TC + NVP, as well as clinical and laboratory safety. Because nevirapine is a strong inducer of hepatic enzymes, pharmacocinetic (PK) assessment will be performed in all patients in the first weeks after switch and 24-hours PK in a subset of 10 patients after 5 days of DTG addition to current regimen, before switching to ABC/3TC/DTG.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed HIV-1 infection (HIV antibody positive confirmation prior to screening)
* Age ≥ 18 years
* Written informed consent
* Male patient or non-pregnant, non-lactating female patient
* On antiretroviral treatment with nevirapine (400 mg per day) plus abacavir/lamivudine for more than 6 months; Nevirapine 400 mg/day being administered as either 1 x 200 mg IR x 2/day or 2 x 200 mg IR qd or 1 x 400 mg XR qd
* No history of prior virologic failure on antiretroviral therapy
* HIV-1 RNA < 50 copies/ml for more than 1 year,
* No major IAS-USA nucleoside reverse transcriptase inhibitors or integrase inhibitors resistance mutations on genotypic testing on last plasma sample with HIV-1 RNA > 500 c/mL (if available)
* HLA-B*5701 negative test
* Subjects covered by Health Insurance

Exclusion Criteria:

* Woman of child-bearing potential without effective contraception method. Pregnant or breastfeeding woman.
* Woman expecting to conceive during the study period
* HIV-2 co-infection
* Any prior exposure to integrase inhibitor(s)
* Plasma HIV-1 RNA > 50 c/mL in the past year
* Creatinine clearance < 60 ml/mn (estimated glomerular filtration rate according to the MDRD equation),
* Alkaline phosphatase, ASAT or ALAT ≥ 5 times the upper limit of the norm (ULN)
* Patient with history of decompensated liver disease
* Any major IAS-USA mutation conferring resistance to one or more of reverse transcriptase or integrase inhibitors on any historical plasma genotype if available. Any previous genotype result is valid, with no time limit, as long as the original test result is documented.
* Mycobacteriosis under treatment
* Malignancy requiring chemotherapy or radiotherapy
* Positive HBs Ag
* HCV infection for which specific treatment is ongoing or planned during the study
* Known hypersensitivity to one of the trial drugs, the metabolites or formulation excipients
* Concomitant therapy with antacids or H2 antagonists
* Contraindicated concomitant treatment
* Anticipated non-compliance with the protocol
* Participation in another clinical trial with an on-going exclusion period at screening
* Subject under legal guardianship or incapacitation
* Subject, who in the opinion of the investigator, is unable to complete the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with plasma HIV-1 RNA < 50 copies/mL at week 12 | Week 12

SECONDARY OUTCOMES:
Percentage of patients with Plasma HIV-1 RNA < 50 copies/ml at W24 | Week 24
Percentage of patients with Plasma HIV-1 RNA < 50 copies/ml at W48 | Week 48
Percentage of patients with undetectable plasma viral load (< 1 copies/ml or signal not detected) at W12 | Week 12
Number of patients with undetectable plasma viral load (< 1 copies/ml or signal not detected) at W24 | Week 24
Number of patients with undetectable plasma viral load (< 1 copies/ml or signal not detected) at W36 | Week 36
Number of patients with undetectable plasma viral load (< 1 copies/ml or signal not detected) at W48 | Week 48
Percentage of patients with adverse event of any Grade over 12 weeks | Week 12
Percentage of patients with adverse event of Grade 3 or 4 over 48 weeks | Week 48
CD4 and CD8 measurement | Week 48
  Changes in CD4 and CD8 counts over 48 weeks
Serum creatinine and GFR (MDRD) measurement | Week 48
  Changes in serum creatinine, and GFR (MDRD) from W2 to W48
Urinary albumine:creatinine ratio measurement | Week 48
  Change in urinary albumine:creatinine ratio over 48 weeks
Fasting lipids measurement | Week 48
  Changes in fasting lipids over 48 weeks
Plasma concentration of NVP between Week 0 (W0) and Week 2 (W2) | Week 2
  The mean plasma concentration of nevirapine is measured between W0 and W2 (D0, W1, W2)
Plasma concentration of dolutegravir between W0 and W12 | Week 12
  The mean plasma concentration of dolutegravir is measured between W0 and W12 (W1, W2, W4, W12)
CD14 and usCRP measurement over 48 weeks | Week 48
  Changes in sCD14 and usCRP over 48 weeks (stored plasma)
Evaluation of patient's satisfaction with HIVTSQs and HIVTSQc questionnaires | Week 48
  Patient's satisfaction, evaluated with self-administered questionnaires HIVTSQs and HIVTSQc
Plasma concentration of DTG on 24h at D0 and Week 2 | Week 2
  24h PK parameters of DTG (D0, after 5 days of combination of ABC/3TC + NVP + DTG) with and without NVP (D14)

CONTACTS AND LOCATIONS:
Overall Officials: François RAFFI, Pr, Study Chair — Nantes University Hospital
Locations (2):
- France (2):
  - La Roche-sur-Yon Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes

REFERENCES:
- [Derived] Dailly E, Allavena C, Gregoire M, Reliquet V, Bouquie R, Billaud E, Hernando H, Bouchez S, Deslandes G, Hall N, Jolliet P, Raffi F. Influence of nevirapine administration on the pharmacokinetics of dolutegravir in patients infected with HIV-1. J Antimicrob Chemother. 2015 Dec;70(12):3307-10. doi: 10.1093/jac/dkv245. Epub 2015 Aug 13. PMID 26271944